CLINICAL TRIAL: NCT02834962
Title: Study of Single And Double Bundle ACL Graft Cross-sectional Dimensions Compared With Native ACL
Brief Title: Study of Single And Double Bundle Anterior Cruciate Ligament (ACL) Graft Cross-sectional Dimensions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Jia-kuo yu, Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACLMRI-1
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Rupture of Anterior Cruciate Ligament
Keywords: Anterior Cruciate Ligament Reconstruction
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- single bundle ACLR (Experimental): patients undergo single bundle ACL reconstruction
  Interventions: Procedure: single bundle ACL reconstruction
- double bundle ACLR (Active Comparator): patients undergo double bundle ACL reconstruction
  Interventions: Procedure: double bundle ACL reconstruction

INTERVENTIONS:
Procedure: single bundle ACL reconstruction — anterior cruciate ligament reconstruction using single bundle technique
  Arms: single bundle ACLR
Procedure: double bundle ACL reconstruction — anterior cruciate ligament reconstruction using double bundle technique
  Arms: double bundle ACLR

SUMMARY:
To study the difference between single and double bundle ACL graft cross-sectional dimensions compared with native ACL using postoperative 3-D MRI.

DETAILED DESCRIPTION:
The investigators divide 100 patients with ACL rupture into 2 groups. Group A undergo single bundle anterior cruciate ligament reconstruction (ACLR). Group B undergo double bundle ACL reconstruction. At 3-6 weeks post operation, all the patients undergo 3-D MRI examination of both knees. The investigators reconstruct 3-D models of reconstructed ACL and native ACL, and compare the difference between single and double bundle graft.

ELIGIBILITY:
Inclusion Criteria:

* ACL rupture patients aged between 10 to 50 years

Exclusion Criteria:

* combined severe injuries to the operated knee (additional ligament rupture, major meniscus loss, patella instability, cartilage damage >2°, pathologic leg axis deviation)
* any injury or surgery to the contralateral knee
* any inflammatory or systemic disease, neuromuscular disease in the lower limbs,any recent knee infection

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
cross-sectional area of the reconstructed ACL | 3-6 weeks
long to short axis ratio of the cross-sectional area of the reconstructed ACL | 3-6 weeks
long axis of the cross-sectional area of the reconstructed ACL | 3-6 weeks
short axis of the cross-sectional area of the reconstructed ACL | 3-6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Kuo Yu, Study Chair — Peking University Third Hospital